CLINICAL TRIAL: NCT04507841
Title: Niraparib for the Neoadjuvant Treatment of Unresectable Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: West China Second University Hospital (Other); Qilu Hospital of Shandong University (Other); Renmin Hospital of Wuhan University (Other); Sun Yat-sen University Cancer Center, Sun Yat-sen University (Unknown); Guangdong Provincial People's Hospital Affiliated to Southern Medical University (Unknown)
Responsible Party: Principal Investigator, Qinglei Gao, Clinical Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-TJ-OVNN
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib group (Experimental): Niraparib was used in patients with newly diagnosed ovarian cancer before any treatment with an individualized starting dose of 200mg/day or 300mg/day based on body weight or platelet count.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Neoadjuvant niraparib monotherapy with an individualized starting dose of 200mg/day or 300mg/day based on body weight or platelet count. The 28-day treatment cycle consists of 21 days of medication followed by a 7-day break. Two cycles of neoadjuvant niraparib monotherapy were used, and the investigator may choose to have an additional cycle based on the patient's condition.

SUMMARY:
This is a prospective, interventional, single-arm, open-label, phase II study to evaluate the safety and efficacy of niraparib monotherapy as neoadjuvant therapy in patients with advanced ovarian cancer, primary peritoneal cancer, fallopian tube cancer ((FIGO stage III or IV), who had low likelihood of achieving R0 cytoreduction by imaging assessment or laparoscopic evaluation, or cannot tolerate PDS by poor conditions.

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent form must be provided before any procedure of the trial, and the informed consent form shall be filed in the research center;
2. Female patients aged between 18 and 75 years old;
3. Patients received open surgery, laparoscopic surgery, or coarse needle aspiration biopsy and confirmed as high-grade serous or endometrioid ovarian cancer, peritoneal cancer, or fallopian tube cancer (hereinafter referred to as ovarian cancer). FIGO stage III-IV;
4. BRCA1/2 gene mutation or HRD was confirmed by tissue or blood samples detected by the testing institution designated by the research center;
5. Blood and tissue samples can be obtained before, during, and after treatment, and the subjects agree to submit the blood and tissue samples to the central laboratory for the expanded research purposes of the trial, including but not limited to: I. possible gene-related research. II. Possible tumor markers related studies;
6. There is at least one lesion that can be measured by CT / MRI;
7. The professional gynecological oncologists appointed by each center should judge the patients who can not achieve R0 tumor reduction or can not tolerate surgery,

   The criteria for failure to achieve R0 tumor reduction include but are not limited to:

   i. Fagotti score ≥ 8 [2];

   II. When the laparoscopic evaluation method is difficult to implement, the upper abdominal CT Score ≥ 3 can be used [3].

   The criteria for intolerance to surgery can be considered as follows:

   III. advanced age: age ≥ 80;

   IV. body mass index: BMI ≥ 40.0;

   v. A variety of chronic diseases;

   Vi. malnutrition or hypoproteinemia;

   VII. Moderate to massive ascites;

   VIII. Newly diagnosed venous thromboembolism;

   IX. physical status: ECOG > 2.
8. The expected survival time was more than 12 weeks;
9. The ECOG score was 0-2;
10. Good organ function, including:

    i. Bone marrow function: neutrophil count ≥ 1500 / μ L; platelet ≥ 100000 / μ L; hemoglobin ≥ 10g / dl

    II. Liver function: total bilirubin ≤ 1.5 times of the upper limit of normal value or direct bilirubin ≤ 1.0 times of the upper limit of normal value; AST and alt ≤ 2.5 times of the upper limit of normal value; when liver metastasis exists, it must be ≤ 5 times of the upper limit of normal value

    III. renal function: serum creatinine ≤ 1.5 times the upper limit of normal value, or creatinine clearance rate ≥ 60ml / min (calculated according to Cockcroft Gault formula);
11. For women with fertility potential, if blood test or urine pregnancy test is negative within one week before enrollment, effective contraceptive measures must be taken, such as physical barrier contraceptive method (condom) or complete abstinence. Oral, injectable or implantable hormonal contraceptives are not allowed. Or women without reproductive potential, defined as:

    i. Natural menopause and menopause for more than 1 year;

    II. Surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy);

    III. serum follicle-stimulating hormone, luteinizing hormone, and plasma estradiol levels were within the menopausal criteria of the research center laboratory.
12. Understand the trial process and have the ability to comply with the trial protocol for the trial duration, including any treatment, examination, inspection, follow-up, and questionnaire required for the completion of the experiment;
13. The patients were willing to complete the questionnaire survey of quality of life during the trial treatment and follow-up, and agreed that the results of the questionnaire survey could be used in clinical research;
14. The toxicity of any previous chemotherapy has returned to ≤ CTCAE 1 or baseline level, except for sensory neuropathy or alopecia with stable symptoms ≤ CTCAE grade 2.

Exclusion Criteria:

-

The enrolled patients should not contain any of the following conditions:

1. Personnel involved in the formulation or implementation of the research plan;
2. Other clinical drug experiments participated in by using other experimental research drugs at the same time as the study;
3. At the same time of this study, other neoadjuvant therapies for cancer should be used, including but not limited to chemotherapy, radiotherapy, immunotherapy, microbial therapy, traditional Chinese medicine treatment, and other experimental therapies;
4. Those who are known to be allergic to niraparib or active or inactive components of drugs with a similar chemical structure to niraparib;
5. Inability to swallow oral drugs and any gastrointestinal diseases that may interfere with the absorption and metabolism of the study drugs, such as uncontrollable nausea and vomiting, gastrointestinal obstruction or malabsorption;
6. Have received any anti-cancer treatment for ovarian cancer;
7. Have been treated with known or possible PARP inhibitors in the past;
8. Symptomatic or uncontrolled brain metastases requiring simultaneous treatment, including but not limited to surgery, radiation and / or corticosteroids, or clinical manifestations of spinal cord compression;
9. Major surgery was performed within 3 weeks before the start of the study or did not recover after the operation;
10. The subjects had other malignant diseases in the past 3 years, except skin squamous cell carcinoma, basal-like carcinoma, breast intraductal carcinoma in situ, or cervical carcinoma in situ.
11. The patient had a previous or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
12. Patients with serious and uncontrollable diseases or the general situation of the subjects judged by the researchers to be unsuitable for joining the study, including but not limited to: active viral infection, such as human immunodeficiency virus, hepatitis B, hepatitis C, etc.; severe cardiovascular disease, uncontrollable ventricular arrhythmia, myocardial infarction in the last three months; uncontrollable epileptic grand mal seizure, no control Stable spinal cord compression, superior vena cava syndrome or other mental disorders that affect patients' informed consent; hypertension beyond drug control; immune deficiency (except splenectomy) or other diseases that researchers believe may expose patients to high-risk toxicity; and;
13. Any medical history or existing clinical evidence indicates that there may be confusion of study results, interference with patients' compliance with the trial protocol throughout the study treatment period, or not in the best interests of patients;
14. The patient received platelet or red blood cell transfusion within four weeks before the start of treatment of the study drug;
15. Patients who are pregnant or breastfeeding, or who plan to become pregnant during the study treatment.
16. Unsolved clinical toxicity (≥ grade 2, except alopecia, neuralgia, lymphopenia, and depigmentation of skin)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2023-09-25 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 3-month
  the percentage of patients received R0 resection after Niraparib neoadjuvant treatment.
Overall Response Rate (ORR) After Neoadjuvant treatment | 3-month
  Overall Response Rate according to RECIST1.1 after Neoadjuvant treatment. ORR is defined as the proportion of participants achieving Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST (v.1.1). Per RECIST 1.1, CR is defined as the disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of diameters (SoD) of target lesions.

SECONDARY OUTCOMES:
Disease Control Rate | 3-month
  Disease control rate is defined as the proportion of participants achieving Complete Response (CR), Partial Response (PR) or Stable Disease (SD) according to RECIST1.1 and CA125 according to GCIC guidelines
Complete pathologic response rate | 3-month
  Complete pathologic response rate is measured according to Miller-Panye system.
Progression Free Survival (PFS) | 3-year
  PFS is defined as the time in months from the date of first study drug administration to the date of first documentation of progressive disease (PD) or death as assessed by the Investigator per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Overall survival (OS) | 5-year
  Overall survival. OS is defined as the time from the study enrollment to death due to any cause.
Quality of Life (QOL) measures using Functional Assessment of Cancer Therapy (FACT- ovarian cancer) | 5 years
  To evaluate quality of life (QOL) for the subjects undergoing this treatment, using validated tools. QOL will be assessed every 3 months during treatment course. [Functional Assessment of Cancer Therapy - Ovarian Cancer questionnaire (score range from 0 to 160. Higher scores represent better quality of life.
Patient report outcome, EQ-VAS | 3 years
  life quality assessment. EQ-VAS, EuroQol-visual analogue scales. Score range from 0 [worse outcome] to 10 [better outcome]).
Rate of treatment interruption and termination | 5 years
  The rate of treatment interruption and termination caused by patients' intolerance of treatment side effects and other reasons;
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 5 years
  To further describe safety and assess toxicities encountered with the use of the proposed treatment regimen in patients with stage III, all stage IV ovarian cancer.
Overall Response Rate (ORR) during niraparib maintain treatment | 1 year
  Overall Response Rate according to RECIST1.1 during niraparib maintain treatment.
  ORR is defined as the proportion of participants achieving Complete Response (CR) or Partial Response (PR) as assessed by the investigator per RECIST (v.1.1). Per RECIST 1.1, CR is defined as the disappearance of all target lesions; PR is defined as at least a 30% decrease in the sum of diameters (SoD) of target lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, MD. PhD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Contact Prof. Gao for primary data.

REFERENCES:
- [Background] Mirza MR, Monk BJ, Herrstedt J, Oza AM, Mahner S, Redondo A, Fabbro M, Ledermann JA, Lorusso D, Vergote I, Ben-Baruch NE, Marth C, Madry R, Christensen RD, Berek JS, Dorum A, Tinker AV, du Bois A, Gonzalez-Martin A, Follana P, Benigno B, Rosenberg P, Gilbert L, Rimel BJ, Buscema J, Balser JP, Agarwal S, Matulonis UA; ENGOT-OV16/NOVA Investigators. Niraparib Maintenance Therapy in Platinum-Sensitive, Recurrent Ovarian Cancer. N Engl J Med. 2016 Dec 1;375(22):2154-2164. doi: 10.1056/NEJMoa1611310. Epub 2016 Oct 7. PMID 27717299
- [Background] Gonzalez-Martin A, Pothuri B, Vergote I, DePont Christensen R, Graybill W, Mirza MR, McCormick C, Lorusso D, Hoskins P, Freyer G, Baumann K, Jardon K, Redondo A, Moore RG, Vulsteke C, O'Cearbhaill RE, Lund B, Backes F, Barretina-Ginesta P, Haggerty AF, Rubio-Perez MJ, Shahin MS, Mangili G, Bradley WH, Bruchim I, Sun K, Malinowska IA, Li Y, Gupta D, Monk BJ; PRIMA/ENGOT-OV26/GOG-3012 Investigators. Niraparib in Patients with Newly Diagnosed Advanced Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2391-2402. doi: 10.1056/NEJMoa1910962. Epub 2019 Sep 28. PMID 31562799
- [Background] Berek JS, Matulonis UA, Peen U, Ghatage P, Mahner S, Redondo A, Lesoin A, Colombo N, Vergote I, Rosengarten O, Ledermann J, Pineda M, Ellard S, Sehouli J, Gonzalez-Martin A, Berton-Rigaud D, Madry R, Reinthaller A, Hazard S, Guo W, Mirza MR. Safety and dose modification for patients receiving niraparib. Ann Oncol. 2018 Aug 1;29(8):1784-1792. doi: 10.1093/annonc/mdy181. PMID 29767688
- [Background] Mirza MR, Avall Lundqvist E, Birrer MJ, dePont Christensen R, Nyvang GB, Malander S, Anttila M, Werner TL, Lund B, Lindahl G, Hietanen S, Peen U, Dimoula M, Roed H, Or Knudsen A, Staff S, Krog Vistisen A, Bjorge L, Maenpaa JU; AVANOVA investigators. Niraparib plus bevacizumab versus niraparib alone for platinum-sensitive recurrent ovarian cancer (NSGO-AVANOVA2/ENGOT-ov24): a randomised, phase 2, superiority trial. Lancet Oncol. 2019 Oct;20(10):1409-1419. doi: 10.1016/S1470-2045(19)30515-7. Epub 2019 Aug 29. PMID 31474354
- [Derived] Xia Y, Huang P, Qian YY, Wang Z, Jin N, Li X, Pan W, Wang SY, Jin P, Drokow EK, Li X, Zhang Q, Zhang Z, Li P, Fang Y, Yang XP, Han Z, Gao QL. PARP inhibitors enhance antitumor immune responses by triggering pyroptosis via TNF-caspase 8-GSDMD/E axis in ovarian cancer. J Immunother Cancer. 2024 Oct 4;12(10):e009032. doi: 10.1136/jitc-2024-009032. PMID 39366751
- [Derived] Zhou D, Liu J, Liu R, Li H, Huang Y, Ma D, Hong L, Gao Q. Effectiveness and Safety of Niraparib as Neoadjuvant Therapy in Advanced Ovarian Cancer With Homologous Recombination Deficiency (NANT): Study Protocol for a Prospective, Multicenter, Exploratory, Phase 2, Single-Arm Study. Front Oncol. 2022 Mar 23;12:852772. doi: 10.3389/fonc.2022.852772. eCollection 2022. PMID 35402241